CLINICAL TRIAL: NCT04373590
Title: Mental Healthcare Decision-Making and Decision Support Among Emerging Adults Enrolled in Coordinated Specialty Care for Early Psychosis
Brief Title: Decision-making and Decision Support Among Emerging Adults With First Episode Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Principal Investigator, Yaara Zisman Ilani, Assistant Professor, Temple University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 24734
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Early Psychosis
MeSH Terms: conditions — Psychotic Disorders | interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Randomization is accomplished using a HIPAA-compliant, Internet-based randomization service (studyrandomizer.com) using permuted blocks of 5. Patients and the participating psychiatrist are not blinded to the condition assigned to them; however, they are not given any explicit information on the DA. The psychiatrist was provided with the DA and received information about it as the DA is delivered by the psychiatrist for patients who are randomized to receive it. The RA who recruit and administer assessments to participants is not blinded to condition, except at baseline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decision aid (DA) (Experimental): a one-page DA for use during the psychiatric consultation to help patients and clinicians discuss relevant treatment options pertaining to antipsychotics.
  Interventions: Behavioral: Decision aid
- Treatment as usual (TAU) (No Intervention): Treatment as usual without the DA

INTERVENTIONS:
Behavioral: Decision aid — The chosen intervention is a one-page DA developed by the first author, published and fully described elsewhere (Zisman-Ilani et al., 2017; Zisman et al., 2018) for use during the psychiatric consultation to help patients and clinicians discuss relevant treatment options pertaining to antipsychotics such as medication nonadherence and self-tapering. The DA format is a simple one-page table with rows containing frequently asked questions by patients about their treatment options and the benefits, risks, and implications of differing decisions. The columns display the treatment options available for the treatment decision in question: continuing, adjusting, or discontinuing antipsychotic medications.
  Arms: Decision aid (DA)

SUMMARY:
The purpose of this study is to evaluate the impact of an antipsychotic medication decision aid and interpersonal and cognitive factors, such as attachment style and motivation, on emerging adults' ability to engage in shared decision making regarding their medications.

DETAILED DESCRIPTION:
The long-term occupational, social, and economic outcomes associated with psychosis make it an urgent public health problem. Coordinated specialty care (CSC) is now the gold standard for early psychosis, demonstrating positive clinical and functional effects in the short-term, and longer-term reduced hospitalization rates. These services include an array of treatment options, including psychotropic medications, individual psychotherapy, family education, and support, and occupational therapy and supported employment/education.

While a shorter period between psychosis onset and receipt of appropriate care is associated with better outcomes, emerging adults often experience significant delays before receiving treatment, and a large percentage disengage from services once they are commenced. Decisional conflict about treatment options (i.e., feeling conflicted about which option to choose) and interpersonal factors such as attachment style and trust in health providers can contribute to decision delay and discontinuance of chosen options. Decision support tools (e.g., decision aids), have been shown to reduce decisional conflict as well as improve service engagement. A requisite step in expanding the array of decision support tools available to emerging adults experiencing early psychosis is to better understand their decision-making ability, capacity, and motivation to engage in decision making and how these relate to their engagement in CSC.

It is well recognized that individuals who are being prescribed antipsychotic medications often face decisional conflict about their treatment options. An especially controversial decision is whether individuals should continue taking medication at the same dose or adjust the dose whilst monitoring their symptoms. This dilemma is the result of some uncertainty about the appropriate treatment strategy for long-term management of psychosis. The present project focuses on evaluating the feasibility and effectiveness of the use of a decision aid for making decisions about antipsychotic medication.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 25 years
* Experiencing early psychosis, defined as psychosis lasting 18 months or less between the time when threshold symptom criteria were reached (as determined by the admitting CSC program assessor) and the date of CSC program enrollment
* Planning to attend a medication appointment with a participating CSC psychiatrist
* Ability to speak and understand English
* Ability to provide informed consent as assessed by research staff using procedures discussed by Carpenter et al. (2000) including a demonstrated understanding and recall of study procedures, rather than passive consent, and allowance of repetition of study procedures until there is understanding and recall.

Exclusion Criteria:

* Have a legal guardian
* Have identified co-occurring dementia, delirium, or intellectual disability that will likely affect their ability to provide informed consent or participate in the data collection procedures.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Change in antipsychotics knowledge | Baseline (Pre-appointment interview ) and post appointment interview ( same 1 day of the appointment )
  Scale to assess change in knowledge about antipsychotic medications over time (9 items)
Decision-making self-efficacy | Post appointment interview (1 day of the appointment )
  Decision Self-Efficacy (DSE) scale to assess decision self-efficacy (11 items)
Decision-making attitudes | Post appointment interview (1 day of the appointment )
  Decision Attitude Scale (DAS) to assess decision-making attitudes (10 items)
Decisional Conflict | Post appointment interview (1 day of the appointment )
  Decisional Conflict Scale (DCS) to assess level of decisional conflict (15 items)
Shared decision making | Post appointment interview (1 day of the appointment )
  collaboRATE scale to assess level of shared decision making after an appointment (3 items)
Change in medication adherence | Baseline (Pre-appointment interview ) and post appointment interview ( same 1 day of the appointment ), 3 months follow-up , 6 months follow-up .
  Brief Adherence Rating Scale (BARS) to assess change in medication adherence over time (8 items)
Change in service use | Baseline (Pre-appointment interview ) and post appointment interview ( same 1 day of the appointment ), 3 months follow-up , 6 months follow-up .
  Service Use and Resource Form for Monthly Items (SURF-M) scale to assess change in service use over time (66 items)
Service engagement | Baseline (Pre-appointment interview )
  Service Engagement Scale (SES) to assess level of service engagement (14 items)

SECONDARY OUTCOMES:
Apathy | Baseline (Pre-appointment interview )
  Marin Apathy Evaluation Scale to assess apathy (18 items)
Attachment style | Baseline (Pre-appointment interview )
  Experiences in Close Relationships-Revised (ECR-R) Questionnaire to assess attachment style (36 items)
Working alliance | Baseline (Pre-appointment interview )
  Working Alliance Inventory (WAI) to assess alliance (36)
Trust | Baseline (Pre-appointment interview )
  Trust in the Medical Profession Scale to assess level of trust in the clinician (11 items)
Cognitive functioning | Baseline (Pre-appointment interview )
  Brief Assessment of Cognition in Schizophrenia (BACS) - a battery to assess aspects of cognition such as verbal memory and attention.
Insight | Baseline (Pre-appointment interview )
  Birchwood Insight Scale to assess insight to the illness (8 items)
Self-stigma | Baseline (Pre-appointment interview )
  Internalized Stigma of Mental Illness (ISMI) Scale - Brief Version, to assess mental health self-stigma (10 items)

CONTACTS AND LOCATIONS:
Locations (1):
- Psychosis Education, Assessment, Care and Empowerment (PEACE), Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zisman-Ilani Y, Shern D, Deegan P, Kreyenbuhl J, Dixon L, Drake R, Torrey W, Mishra M, Gorbenko K, Elwyn G. Continue, adjust, or stop antipsychotic medication: developing and user testing an encounter decision aid for people with first-episode and long-term psychosis. BMC Psychiatry. 2018 May 22;18(1):142. doi: 10.1186/s12888-018-1707-x. PMID 29788933
- [Derived] Zisman-Ilani Y, Hurford I, Bowen A, Salzer M, Thomas EC. Evaluating the feasibility of a decision aid to promote shared decision making among young adults with first-episode psychosis: protocol for a pilot study. Pilot Feasibility Stud. 2021 Jan 11;7(1):22. doi: 10.1186/s40814-020-00757-0. PMID 33431018